CLINICAL TRIAL: NCT04813562
Title: A Single-center, Randomized, Double Blinded, Placebo Controlled, Phase 2 Clinical Trial of Recombinant COVID-19 Vaccine (CHO Cells), in the Subjects From Healthy Aged 18 Years and Above
Brief Title: Immunogenicity and Safety of Recombinant COVID-19 Vaccine (CHO Cells)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Academy of Military Medical Sciences，Academy of Military Sciences，PLA ZHONGYIANKE Biotech Co, Ltd. LIAONINGMAOKANGYUAN Biotech Co, Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JSVCT097
Record Dates: First submitted 2021-03-19; First posted 2021-03-24 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
Keywords: Immunogenicity; Safety; COVID-19 vaccine; Recombinant vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Middle-dose vaccine (18-59 years) (Experimental): Three doses of middle-dose experimental vaccine at the schedule of day 0, 28, 56
  Interventions: Biological: a middle-dose recombinant COVID-19 vaccine (CHO Cell) (18-59 years) at the schedule of day 0, 28, 56
- High-dose vaccine (18-59 years) (Experimental): Two doses of High-dose vaccine at the schedule of day 0, 28, 56
  Interventions: Biological: a high-dose recombinant COVID-19 vaccine (CHO Cell) (18-59 years) at the schedule of day 0, 28, 56
- Middle-dose vaccine (60-85 years) (Experimental): Three doses of middle-dose experimental vaccine at the schedule of day 0, 28, 56
  Interventions: Biological: a middle-dose recombinant COVID-19 vaccine (CHO Cell) (60-85 years) at the schedule of day 0, 28, 56
- High-dose vaccine (60-85 years) (Experimental): Two doses of High-dose experimental vaccine at the schedule of day 0, 28, 56
  Interventions: Biological: a high-dose recombinant COVID-19 vaccine (CHO Cell) (60-85 years) at the schedule of day 0, 28, 56
- Middle-dose placebo (18-59 years) (Placebo Comparator): Three doses of middle-dose placebo at the schedule of day 0, 28, 56
  Interventions: Biological: a middle-dose placebo (18-59 years) at the schedule of day 0, 28, 56
- High-dose placebo (18-59 years) (Placebo Comparator): Two doses of High-dose placebo at the schedule of day 0, 28, 56
  Interventions: Biological: a high-dose placebo (18-59 years) at the schedule of day 0, 28, 56
- Middle-dose placebo (60-85 years) (Placebo Comparator): Three doses of middle-dose placebo at the schedule of day 0, 28, 56
  Interventions: Biological: a middle-dose placebo (60-85 years) at the schedule of day 0, 28, 56
- High-dose placebo (60-85 years) (Placebo Comparator): Two doses of High-dose placebo at the schedule of day 0, 28, 56
  Interventions: Biological: a high-dose placebo (60-85 years) at the schedule of day 0, 28, 56

INTERVENTIONS:
Biological: a middle-dose recombinant COVID-19 vaccine (CHO Cell) (18-59 years) at the schedule of day 0, 28, 56 — 18-59 years,Three doses of middle-dose (20µg/0.5ml) recombinant COVID-19 vaccine (CHO Cell) at the schedule of day 0, 28, 56.
  Arms: Middle-dose vaccine (18-59 years)
Biological: a high-dose recombinant COVID-19 vaccine (CHO Cell) (18-59 years) at the schedule of day 0, 28, 56 — 18-59 years,Three doses of high-dose (40µg/0.5ml) recombinant COVID-19 vaccine (CHO Cell) at the schedule of day 0, 28, 56.
  Arms: High-dose vaccine (18-59 years)
Biological: a middle-dose recombinant COVID-19 vaccine (CHO Cell) (60-85 years) at the schedule of day 0, 28, 56 — 60-85 years,Three doses of middle-dose (20µg/0.5ml) recombinant COVID-19 vaccine (CHO Cell) at the schedule of day 0, 28, 56.
  Arms: Middle-dose vaccine (60-85 years)
Biological: a high-dose recombinant COVID-19 vaccine (CHO Cell) (60-85 years) at the schedule of day 0, 28, 56 — 60-85 years,Three doses of high-dose (40µg/0.5ml) recombinant COVID-19 vaccine (CHO Cell) at the schedule of day 0, 28, 56.
  Arms: High-dose vaccine (60-85 years)
Biological: a middle-dose placebo (18-59 years) at the schedule of day 0, 28, 56 — 18-59 years,Three doses of middle-dose (0.5ml) placebo at the schedule of day 0, 28, 56.
  Arms: Middle-dose placebo (18-59 years)
Biological: a high-dose placebo (18-59 years) at the schedule of day 0, 28, 56 — 18-59 years,Three doses of high-dose (0.5ml) placebo at the schedule of day 0, 28, 56.
  Arms: High-dose placebo (18-59 years)
Biological: a middle-dose placebo (60-85 years) at the schedule of day 0, 28, 56 — 60-85 years,Three doses of middle-dose (0.5ml) placebo at the schedule of day 0, 28, 56.
  Arms: Middle-dose placebo (60-85 years)
Biological: a high-dose placebo (60-85 years) at the schedule of day 0, 28, 56 — 60-85 years,Three doses of high-dose (0.5ml) placebo at the schedule of day 0, 28, 56.
  Arms: High-dose placebo (60-85 years)

SUMMARY:
This is a phase Ⅱ, randomized, placebo-controlled, double-blind study, to evaluate immunogenicity and safety of a recombinant COVID-19 vaccine (CHO cells) in the subjects from healthy adults and elderly adults aged 18 years and above (aged 18-60 and 60-85 years) with an immunization procedure (0, 28, 56 days).

DETAILED DESCRIPTION:
This is a phase Ⅱ, single-center, randomized, double-blind, placebo-controlled study, to evaluate the immunogenicity and safety of the recombinant COVID-19 vaccine (CHO cells) in the subjects from healthy adults and elderly adults aged 18 years and above (aged 18-60 and 60-85 years) . The phase Ⅱ clinical trials designed 4 research group, including an immunization procedures (0, 28, 56 days), two doses (20μg/0.5ml, 40μg/0.5ml) and two ages group (adults and elder): Each group including 120 participants. Vaccination or placebo group will be randomly assigned to receive in a 5:1 ratio, 480 in total.

Cellular immune blood samples were collected from the top 96 subjects (i.e., the top 24 in each study group, vaccine group: control group =5:1), and Elispot test and cytokine staining (ICS)/flow assay were performed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects of ≥ 18 years old.
* The subject can understand and voluntarily sign the informed consent.
* Axillary temperature ≤37.0℃.
* General good health as established by medical history and physical examination

Exclusion Criteria:

* Have a history of close contact with a confirmed case of SARS-CoV-2, an asymptomatic infection in the previous 14 days, or a travel history/residential history in a community where a case has been reported.
* Have a history of contact with a person infected with SARS-CoV-2(a person with a positive nucleic acid test) in the previous 14 days.
* Patients with fever or respiratory symptoms who have been to middle or high-risk areas in the past 14 days or have exit history, or come from communities with case reports.
* In the past 14 days, there have been 2 or more cases of fever and/or respiratory symptoms in small areas such as homes, offices, school classes, etc.
* Have a history of SARS.
* Have a history of SARS-CoV-2 infection or history of Coronavirus Vaccination (including Emergency Vaccine and Experimental Vaccine).
* Positive in SARS-CoV-2 IgG or IgM antibody screening.
* Have a history of HIV infection;
* Women who are breastfeeding, pregnant, or planning to become pregnant during 6 months after full-course vaccination (based on the subject's self-report and blood pregnancy test results for women of childbearing age).
* Have a history of asthma, a history of vaccine or vaccine component allergy, have serious adverse reactions to the vaccine, such as urticaria, dyspnea, angioedema.
* Subjects with congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.
* Subjects with autoimmune diseases or immunodeficiency/immunosuppression.
* Subjects with severe chronic diseases, severe cardiovascular diseases, hypertension(sbp≥160mmHg and/or dbp≥100mmHg) and diabetes that cannot be controlled by drugs, liver and kidney diseases, malignant tumors, etc.
* Subjects with severe neurological disease (epilepsy, convulsions or convulsions) or mental illness.
* Subjects with thyroid disease or history of thyroidectomy, no spleen, functional asthenia, and any spleen or splenectomy caused by any condition.
* Abnormal blood coagulation function diagnosed by a doctor (such as coagulation factor deficiency, coagulopathy, abnormal platelet) or obvious bruise or coagulation disorder.
* Have received immunosuppressant therapy, cytotoxic therapy, and inhaled corticosteroids in the past 6 months (excluding corticosteroid spray therapy for allergic rhinitis and surface corticosteroid therapy for acute non-complicated dermatitis).
* Received blood products within 3 months before receiving trial vaccine.
* Received other study drugs within 30 days before receiving the trail vaccine.
* Received a live attenuated vaccine within 14 days before receiving the experimental vaccine.
* Received a subunit or inactivated vaccine within 7 days before receiving the experimental vaccine.
* Various acute or chronic diseases occurred in the past 7 days.
* Have a long history of alcohol or drug abuse.
* Had urticaria one year before receiving the experimental vaccine;
* congenital or acquired angioedema/neuroedema;
* According to the judgment of the investigator, the subject has any other factors that are not suitable for participating in the clinical trial, or Or influence the subject to sign the informed consent.

Exclusion criteria of subsequent dose:

* Patients with severe allergic reactions after the previous dose of vaccination;
* Patients with serious adverse reactions causally related to the previous dose of vaccination.
* For those newly discovered or newly discovered after the first vaccination that does not meet the first-dose selection criteria or meets the first-dose exclusion criteria, the investigator will determine whether to continue participating in the study.
* Other exclusion reasons suggested by the researchers.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2021-03-23 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
The positive conversion rate of anti-SARS-CoV-2 specific neutralizing antibody (eucivirus neutralization assays) | 30 days after full-course vaccination in each study group
The incidence of adverse reaction (AR) | 0 to 7 days after vaccination in each study group

SECONDARY OUTCOMES:
The incidence of adverse events (AE) | 0 to 30 days after vaccination in each study group
The incidence of severe adverse events (SAE) | 12 months after prime and boost vaccination
The Geometric mean titer (GMT) of anti-SARS-CoV-2 specific neutralizing antibody (euvirus and pseudovirus neutralization assays) | 14 days, 30 days, 6 months and 12 months after full-course vaccination in each study group
The Geometric mean fold increase (GMI) of anti-SARS-CoV-2 specific neutralizing antibody (euvirus and pseudovirus neutralization assays) | 14 days, 30 days, 6 months and 12 months after full-course vaccination in each study group
The positive conversion rate of anti-SARS-CoV-2 specific neutralizing antibody (eucivirus neutralization assays) | 14 days, 6 months and 12 months after full-course vaccination in each study group
The positive conversion rate of anti-SARS-CoV-2 specific neutralizing antibody (pseudovirus neutralization assays) | 14 days, 30days, 6 months and 12 months after full-course vaccination in each study group
The positive conversion rate of the SARS-CoV-2 neutralizing antibody and the S-RBD protein specific antibody | 14 days, 30days, 6 months and 12 months after full-course vaccination in each study group
The GMT of the SARS-CoV-2 neutralizing antibody and the S-RBD protein specific antibody | 14 days, 30days, 6 months and 12 months after full-course vaccination in each study group
The GMI of the SARS-CoV-2 neutralizing antibody and the S-RBD protein specific antibody | 14 days, 30days, 6 months and 12 months after full-course vaccination in each study group

OTHER OUTCOMES:
The geometric mean titer (GMT) ratio of the SARS-CoV-2 neutralizing antibody and the S-RBD protein specific antibody in each study groups | 14 days, 30days, 6 months and 12 months after full-course vaccination in each study group
Subtypes of IgG antibodies against the S-RBD protein of SARS-CoV-2 after immunization in each study group | 14 days, 30days, 6 months and 12 months after full-course vaccination in each study group
The proportion of IFN-γ secreted by T cells at Day 14 using ELISpot detection method | Day 14 after full-course vaccination in each study group
The Intracellular cytokine staining (ICS)/flow cytometry was used to detect the Th1/Th2 immune response after immunization (CD3+/CD4+/CD8+ T cells, and cytokines TNFα/IFNγ/IL2/IL4). | Day 14 after full-course vaccination in each study group

CONTACTS AND LOCATIONS:
Overall Officials: Fengcai Zhu, Doctor, Principal Investigator — Jiangsu Provincial Center for Disease Control and Prevention
Locations (1):
- Jiangsu Provincial Center for Diseases Control and Prevention, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Luo D, Pan H, He P, Yang X, Li T, Ning N, Fang X, Yu W, Wei M, Gao H, Wang X, Gu H, Mei M, Li X, Zhang L, Li D, Gao C, Gao J, Fei G, Li Y, Yang Y, Xu Y, Wei W, Sun Y, Zhu F, Hu Z, Wang H. A randomized, double-blind, placebo-controlled phase 1 and phase 2 clinical trial to evaluate efficacy and safety of a SARS-CoV-2 vaccine SCoK in adults. Clin Transl Med. 2022 Sep;12(9):e1016. doi: 10.1002/ctm2.1016. PMID 36103390